CLINICAL TRIAL: NCT02205242
Title: BACE Trial - Physical Activity as a Crucial Patient Reported Outcome in COPD
Brief Title: BACE Trial Substudy 1 - PROactive Substudy
Acronym: PROactive
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wim Janssens (Other)
Collaborators: Pro-Active Medical Pty Ltd (Industry)
Responsible Party: Sponsor-Investigator, Wim Janssens, MD. Phd., KU Leuven
Organization: KU Leuven (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: s55829 - PROactive Substudy
Record Dates: First submitted 2014-07-22; First posted 2014-07-31 (Estimated); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: AECOPD; Chronic Obstructive Pulmonary Disease; Acute exacerbation; Hospitalization; Azithromycin; Macrolides; Randomized Controlled Trial; Placebo; Physical Activity; PRO-Active; Activity Monitor
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Azithromycin; Fitness Trackers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azithromycin (Experimental): N = 250 From day 1 up to and including day 3: 500 mg azithromycin PO once a day From day 4 up to and including day 90: 250 mg azithromycin PO once every 2 days
  N= 30 During 7 days post discharge from hospital (0 months), 3 months and 9 months, the patient will wear the Dynaport® which will register the patient's physical activity
  Interventions: Drug: Azithromycin; Device: Dynaport®
- Placebo (Placebo Comparator): N = 250 From day 1 up to and including day 3: 500 mg placebo PO once a day From day 4 up to and including day 90: 250 mg placebo PO once every 2 days
  N= 30 During 7 days post discharge from hospital (0 months), 3 months and 9 months, the patient will wear the Dynaport® which will register the patient's physical activity
  Interventions: Device: Dynaport®; Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — From day 1 up to and including day 3: 500 mg azithromycin or placebo PO once a day From day 4 up to and including day 90: 250 mg azithromycin or placebo PO once every 2 days
  Other Names: Azitromcyine CF; ATC code: J01FA10
  Arms: Azithromycin
Device: Dynaport® — Registering physical activity during 7 days post discharge from hospital (0 months), 3 months and 9 months
  Other Names: Activity monitor
Drug: Placebo
  Other Names: Inactive substance
  Arms: Placebo

SUMMARY:
A first sub-analysis of the BACE trial will address physical activity levels in a subgroup of the intervention study with portable validated activity monitors.

DETAILED DESCRIPTION:
Physical activity is strongly reduced with exacerbations and failure to increase physical activity is associated with relapse. In addition, physical inactivity is known to be associated with cardiovascular and metabolic morbidity and is one of the strongest predictors of mortality in COPD. Apart from potential direct effects of the intervention on treatment failure and symptoms, positive effects on physical activity may offer considerable benefits in the long run.

Randomized patients that are willing to participate in the sub-study will be monitored for activity by validated and easy-to-wear portable devices (Dynaport®). This activity monitor was recently thoroughly validated for use in COPD by the Pro-Active consortium and will be used at the baseline, 3 months and 9 months visit. We hypothesize that with a positive medical intervention, differences in recovery of physical activity will be appreciated.

Patients will follow the standard protocol but will also wear the activity monitor for 7 days post discharge from hospital (at investigator discretion), at day 90 (end of treatment) and at day 270 (end of follow-up). This device is not only registering physical activity for 7 days but is also coupled to a standardized and patient-validated questionnaire on physical activities which needs to be filled out at day 8 to cover a recall period of 7 (monitored) days.

Patient will have to give informed consent for the additional measures that are related to the activity sub-study. However, individual patients can still opt out for these tests (sub-study) and only participate in the medical intervention study (main study).

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of COPD by medical doctor (based on clinical history OR pulmonary function test)
* Smoking history of at least 10 pack-years (10 pack-years are defined as 20 cigarettes a day for 10 years, or 10 cigarettes a day for 20 years, etc.)
* Current hospitalization for potential infectious AECOPD treated with standard therapy
* History of at least one exacerbation during the last year (prior to the current hospital admission) for which systemic steroids and/or antibiotics were taken
* ECG at admission

Exclusion Criteria:

* Mechanical or non-invasive ventilation at moment of randomization (D1)
* Long QT interval on ECG (QTc > 450msec for males or > 470msec for females)
* History of life-threatening arrhythmias
* Myocardial infarction (NSTEMI or STEMI) less than 6 weeks before start of study drug
* Unstable angina pectoris or acute myocardial infarction (NSTEMI or STEMI) at admission
* Drugs with high risk for long QT interval and torsade de pointes (amiodarone, flecainide, procainamide, sotalol, droperidol, haldol, citalopram, other macrolides)
* Documented uncorrected severe hypokalemia (K+ < 3.0 mmol/L) or hypomagnesemia (Mg2+ < 0.5 mmol/L)
* Chronic systemic steroids (> 4 mg methylprednisolone /day for ≥ 2 months)
* Actual use of macrolides for at least 2 weeks
* Allergy to macrolides
* Active cancer treatment
* Life expectancy < 3 months
* Pregnant or breast-feeding subjects. Woman of childbearing potential must have a pregnancy test performed and a negative result must be documented before start of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-09; Primary Completion 2018-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Difference in Physical Activity (total amount of steps) registered by the Dynaport® during 7 days between discharge from hospital (0 months) and 3 months after randomisation | At discharge from hospital (0 months) and 3 months after start study drug intake
  Physical activity will be quantified as Total amount of steps

SECONDARY OUTCOMES:
Key secondary endpoint: Different change in physical activity (total amount of steps) at 3 months between placebo and azithromycin arm | 0 and 3 months
  Difference between placebo and azithromycin arm in physical activity changes registered by the Dynaport® during 7 days at discharge from hospital (0 months) and at 3 months
Different change in physical activity (total amount of steps) at 9 months between placebo and azithromycin arm | at baseline and 9 months
  Difference between placebo and azithromycin arm in physical activity changes registered by the Dynaport® during 7 days at discharge from hospital (0 months) and at 9 months
Difference in Physical Activity (TSMVA) registered by the Dynaport® during 7 days between discharge from hospital (0 months) and 9 months, or between 3 months and 9 months after randomisation | baseline, 3 and 9 months
  Physical activity will be specified for:
  1. Total amount of steps
  2. Total time spent in moderate to intense physical activity
  3. Sedentary Time (Lying-Sitting) and Time Active (Standing-Locomotion-Shuffeling)
Difference in Physical Activity (TSMVA) registered by the Dynaport® during 7 days between discharge from hospital (0 months) and 3 months after randomisation | At discharge from hospital (0 months) and 3 months after start study drug intake
  Physical activity will be specified for:
  1. Total time spent in moderate to intense physical activity
  2. Sedentary Time (Lying-Sitting) and Time Active (Standing-Locomotion-Shuffeling)

OTHER OUTCOMES:
Exploratory endpoint: sensitivity analysis of primary and secondary endpoints in subgroups | at 0, 3 and 9 months
  * Male vs female
  * Smoker vs ex-smoker (stopped smoking > 6 months)
  * GOLD A, B vs GOLD C vs GOLD D
  * Former GOLD I, II vs III vs IV
  * High CRP (> 50 mg/dL) vs low CRP (< 50 mg/dL)
  * Age < 60 years vs age 60 - 70 years vs age > 70 years
  * Anthonissen I vs Anthonissen II vs Anthonissen III at admission
  * ICS use vs no ICS use

CONTACTS AND LOCATIONS:
Overall Officials: Wim Janssens, MD PhD, Principal Investigator — KU Leuven
Locations (6):
- Belgium (6):
  - St. Pieterziekenhuis, Brussels, Brussels Capital
  - ZNA Middelheim, Antwerp, Flanders
  - Imelda Ziekenhuis, Bonheiden, Flanders
  - UZ Gent, Ghent, Flanders
  - Jessa Ziekenhuis, Hasselt, Flanders
  - UZ Gasthuisberg, Leuven, Flanders

IPD SHARING:
Plan to Share IPD: No